CLINICAL TRIAL: NCT00809757
Title: A Safety, Efficacy, and Tolerability Study of Daily Dosing With Levalbuterol Tartrate HFA MDI and Placebo in Subjects Aged Birth to <48 Months With Asthma
Brief Title: A Safety, Efficacy and Tolerability Study in Pediatric Subjects With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 051-359
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Levalbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 90 ug Levalbuterol (2 actuations)
  Interventions: Drug: Levalbuterol
- 2 (Active Comparator): 0.31 ug Levalbuterol UDV TID
  Interventions: Drug: Levalbuterol UDV TID
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levalbuterol — 90 ug Levalbuterol (2 actuations)
  Other Names: Xopenex HFA Inhalation Aerosol
  Arms: 1
Drug: Levalbuterol UDV TID — 0.31 ug Levalbuterol UDV TID
  Other Names: Xopenex Inhalation Solution
  Arms: 2
Drug: Placebo — Placebo (2 actuations)
  Arms: 3

SUMMARY:
A Safety, Efficacy, and Tolerability Study of Daily Dosing with Levalbuterol Tartrate HFA MDI and Placebo in Subjects Aged Birth to <48 Months with Asthma.

DETAILED DESCRIPTION:
This is a modified-blind, randomized, placebo-controlled, multicenter, parallel-group trial of levalbuterol HFA MDI administered using a facemask and holding chamber in subjects birth to <48 months with asthma. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent/legal guardian must give written informed consent, including privacy authorization, prior to study participation. Complete documentation regarding the consent process must be recorded in the case report form (CRF) and source documentation.
* Subject's parent/legal guardian must be willing and able to comply with the study procedures and visit schedules.
* Subject, male or female, must be between the ages of birth and <48 months, exclusive, at the time of consent.
* Subjects 24 to <48 months of age must have a history of physician-diagnosed asthma (defined as at least 3 episodes of respiratory symptoms consistent with asthma symptoms including, but not limited to, cough, wheeze, or dyspnea).
* Subjects 0 to <24 months of age must have a history of 3 episodes of respiratory symptoms that in the judgement of the investigator could be consistent with asthma or reactive airways disease.
* Subject must be in good health and not affected by any other chronic conditions, including respiratory disorders other than asthma.
* In subjects with a chest radiograph (taken 12 months prior to screening visit), no evidence of any chronic cardiopulmonary condition other than asthma should be present as discerned by the Investigator.
* Subject's parent/legal guardian must be able to complete the diary cards and medical event calendars (MEC) reliably on a daily basis and understand dosing instructions and questionnaire completion.

Exclusion Criteria:

* Subject who requires or is expected to require any disallowed medications
* Subject who has participated in an investigational drug study within 30 days prior to screening, or who is currently participating in another clinical trial.
* Subject or parent/legal guardian who has daily commitments during the study that would interfere with trial measurements, compliance, or both.
* Subject who has a history of hospitalization for asthma, reactive airways disease, or bronchospasm within 4 weeks prior to screening or who is scheduled for in-patient hospitalization, including elective surgery during the course of the trial.
* Subject who has experienced significant blood loss within 60 days of study drug.
* Subject with a clinical diagnosis of cystic fibrosis.
* Subject who was born prematurely, defined as less than 38 weeks gestational age at birth, and is <1 year of age at screening
* Subject whose body weight is less than 7.0 kg at screening. This minimum weight requirement is based upon standard pediatric growth charts [CDC 2000].
* Subject with a known sensitivity to levalbuterol or racemic albuterol, or any of the excipients contained in any of these formulations.
* Subject using any prescription drug with which levalbuterol or racemic albuterol sulfate administration is contraindicated.
* Subject with a history of life-threatening asthma, defined as previous asthma episodes requiring intubation or associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* Subject with clinically significant abnormalities that may interfere with the metabolism or excretion of the study drugs or study participation (eg, abnormalities of renal, hepatic, metabolic, or endocrine function).
* Subject with a history of cancer.
* Subject with any chronic or congenital cardiorespiratory condition other than asthma including, but not limited to, bronchopulmonary dysplasia, congenital heart disease, and cystic fibrosis.
* Subject affected by an upper or lower respiratory tract infection in the 3 weeks prior to screening.
* Subject with a history of ventilation for a respiratory condition occurring at or near birth, including those associated with prematurity or bronchopulmonary dysplasia. Ventilatory support for elective non-cardiopulmonary surgery is not exclusionary. - Subject with any clinically significant abnormal laboratory values (hematology, blood chemistry).
* Subject with a clinically significant abnormal 12-lead ECG that would put the subject at risk for experiencing adverse cardiac effects.
* Subject who is a relative of a staff member.

Max Age: 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (46):
- United States (46):
  - Little Rock Allergy & Asthma Clinical Research Center, Little Rock, Arkansas
  - West Coast Clinical Trials, LLC, Cypress, California
  - Allergy & Asthma Care Center of Southern California, Long Beach, California
  - Clinical Trials of Orange County, Inc., Orange, California
  - Allergy and Asthma Consultants, Redwood City, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - All Seasons Allergy and Asthma Center, P.A., Fort Walton Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Brookstone Centre Parkway, Columbus, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Northern Illinois Research Associates, DeKalb, Illinois
  - Sneeze, Wheeze & Itch Associates LLC, Normal, Illinois
  - Nassim, McMonigle, Mescia & Associates, New Albany, Indiana
  - Grand Blanc Medical, Grand Blanc, Michigan
  - Craig A. Spiegel MD, Bridgeton, Missouri
  - Midwest Allergy and Asthma center, Omaha, Nebraska
  - The Asthma & Allergy Center, P.C., Papillion, Nebraska
  - Maimonides Medical Center, Brooklyn, New York
  - St. Elizabeth Health Center, Utica, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Allergy, Asthma and clinical Research Center, Oklahoma City, Oklahoma
  - Eminence Research, LLC, Oklahoma City, Oklahoma
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - National Allergy, Asthma, and Uticaria Centers, Charleston, South Carolina
  - AAC Research - PC, Charleston, South Carolina
  - ADAC Research, PA, Greenville, South Carolina
  - The Asthma Institute, PLLC, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Isis Clinical Research, LLC, Austin, Texas
  - Sirius Clinical Research, LLC, Austin, Texas
  - Hill Country Family Medical Center, Boerne, Texas
  - TTS Research, Boerne, Texas
  - Allergy/Immunology Research Center of North Texas, Dallas, Texas
  - Dallas Allergy Immunology Research, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Breath of Life Research Institute, Katy, Texas
  - Live Oak Allergy and Asthma Clinic, Live Oak, Texas
  - Quality Assurance Research Center, Inc., San Antonio, Texas
  - Southwest Allergy and Asthma, P.A., San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy & Asthma Care of Waco, Waco, Texas
  - Allergy and Asthma Research Institute, Waco, Texas
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Colonial Heights Pediatrics, Colonial Heights, Virginia
  - Bellingham Asthma, Allergy, & Immunology Clinic, Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Levalbuterol MDI: 90 ug Levalbuterol (2 actuations)
  Levalbuterol: 90 ug Levalbuterol (2 actuations)
- Levalbuterol UDV: 0.31 ug Levalbuterol UDV TID
  Levalbuterol UDV TID: 0.31 ug Levalbuterol UDV TID
Period: Overall Study
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Started | 68 | 65 | 64
Completed | 62 | 60 | 53
Not Completed | 6 | 5 | 11
Not completed — Adverse Event | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 3
Not completed — Subject Uncooperative | 1 | 0 | 2
Not completed — Noncompliance with Medication | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject was randomized but not dosed in the Levalbuterol UDV arm.
Groups:
- Placebo: Placebo Placebo MDI TID
- Levalbuterol MDI: Levalbuterol MDI TID
- Levalbuterol UDV: Levalbuterol UDV TID: 0.31 ug Levalbuterol UDV TID
- Total: Total of all reporting groups
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV | Total
Number analyzed (Participants) | 68 | 65 | 63 | 196
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68 | 65 | 63 | 196
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: Months] | 29.2 (12.17) | 29.3 (12.57) | 28.4 (12.48) | 29.0 (12.35)
Age, Customized [Number; unit: participants]
  0 to < 12 months | 9 | 9 | 9 | 27
  0 to < 24 months | 23 | 23 | 22 | 68
  24 to < 48 months | 45 | 42 | 41 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 24 | 88
  Male | 39 | 30 | 39 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 19 | 56
  Not Hispanic or Latino | 52 | 44 | 44 | 140
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 18 | 23 | 24 | 65
  White | 46 | 39 | 36 | 121
  More than one race | 4 | 2 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 68 | 65 | 63 | 196

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit 4 in the Mean Daily Composite Score Based on the Pediatric Asthma Caregiver Assessments (PACA)
Description: The daily composite score is the sum of the scores of 5 domains: Nocturnal Awakenings Due to Wheeze and Cough, Daytime Wheeze, Daytime Cough, Shortness of Breath, and Asthma Symptom Score. A possible score of 0 (no symptoms) to 19 (severe symptoms).
  The mean daily composite score at Visit 4 is defined as the mean of the daily composite scores in the week prior to Visit 4.
Time Frame: Baseline, Visit 4 (Week 4)
Population: Intent-to-Treat Population. Only those subjects who had non-missing data at Week 4 and at Baseline were included. Subjects who discontinued from the study prior to Week 4 are not included in this analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 59 | 54
units on a scale | -1.21 (2.722) | -0.67 (2.092) | -0.52 (2.843)
Statistical Analysis 1: Comparison: Placebo vs Levalbuterol MDI; 195 subjects were randomized in order to achieve 150 subjects completing the study. The sample size was set based on FDA requirements, and was outside of statistical considerations; Test type: Superiority or Other; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-1.412 to 0.342] — Difference is Placebo MDI minus Levalbuterol UDV
Statistical Analysis 2: Comparison: Placebo vs Levalbuterol UDV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.714 to 0.335] — Difference is Levalbuterol UDV minus Levalbuterol MDI
Statistical Analysis 3: Comparison: Levalbuterol MDI vs Levalbuterol UDV; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-1.080 to 0.771] — Difference is Levalbuterol UDV minus Levalbuterol MDI

2. Secondary Outcome: Change From Baseline to Visit 3 in Mean Daily Composite Score Based on the Pediatric Asthma Caregiver Assessment
Description: The daily composite score is the sum of the scores of 5 domains: Nocturnal Awakenings Due to Wheeze and Cough, Daytime Wheeze, Daytime Cough, Shortness of Breath, and Asthma Symptom Score. A possible score of 0 (no symptoms) to 19 (severe symptoms).
  The mean daily composite score at Visit 3 is defined as the mean of the daily composite scores in the 7 days prior to Visit 3.
Time Frame: Baseline, Visit 3 (Week 3)
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: PBO MDI
  Placebo: Placebo (2 actuations) MDI TID
- Levalbuterol MDI: LEV MDI Levalbuterol: 90 ug Levalbuterol (2 actuations) MDI TID
- Levalbuterol UDV: LEV UDV Levalbuterol UDV TID: 0.31 ug Levalbuterol UDV TID
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 65 | 63 | 56
units on a scale | -0.83 (2.913) | -0.28 (2.490) | -0.22 (2.545)

3. Secondary Outcome: Change From Baseline to Visit 2 to Visit 3 in the Mean Daily Composite Score Based on the Pediatric Asthma Caregiver Assessment
Description: The daily composite score is the sum of the scores of 5 domains: Nocturnal Awakenings Due to Wheeze and Cough, Daytime Wheeze, Daytime Cough, Shortness of Breath, and Asthma Symptom Score. A possible score of 0 (no symptoms) to 19 (severe symptoms).
  The mean daily composite score from Visit 2 to Visit 3 is defined as the mean of the daily composite scores from Visit 2 (inclusive) to the day prior to Visit 3.
Time Frame: The days from Visit 2 (inclusive) to the day prior to Visit 3 - approximately 14 days
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Levalbuterol UDV: LEV UDV 0.31 ug Levalbuterol UDV TID
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 68 | 64 | 59
units on a scale | -0.82 (2.417) | -0.25 (2.041) | -0.15 (2.067)

4. Secondary Outcome: Change From Baseline to Visit 3 to Visit 4 in the Mean Daily Composite Score Based on the Pediatric Asthma Caregiver Assessment
Description: The daily composite score is the sum of the scores of 5 domains: Nocturnal Awakenings Due to Wheeze and Cough, Daytime Wheeze, Daytime Cough, Shortness of Breath, and Asthma Symptom Score. A possible score of 0 (no symptoms) to 19 (severe symptoms).
  The mean daily composite score from Visit 3 to Visit 4 is defined as the mean of the daily composite scores from Visit 3 (inclusive) to the day prior to Visit 4.
Time Frame: The days from Visit 3 (inclusive) to the day prior to Visit 4 - approximately 14 days
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 64 | 62 | 57
units on a scale | -1.08 (2.478) | -0.40 (2.285) | -0.52 (2.331)

5. Secondary Outcome: Change From Baseline to Visit 3 in the Mean Daily Composite Score Based on the Daytime and Nighttime Asthma Symptom Scores as Measured by the Pediatric Asthma Questionnaire (PAQ)
Description: The daily composite score is the sum of the scores of 7 items: Difficulty Breathing, Cough, Wheeze, Activity Limitation, Level of Activity Limitation, Overall Symptom Score, and Nighttime Asthma. The range for the PAQ is 0 (no symptoms) to 27 (severe symptoms).
  The mean daily composite score at Visit 3 is defined as the mean daily composite scores for 7 days prior to Visit 3.
Time Frame: Baseline, Visit 3 (Week 3)
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 65 | 63 | 56
units on a scale | -0.82 (3.457) | -0.45 (3.522) | 0.00 (3.199)

6. Secondary Outcome: Change From Baseline to Visit 4 in the Mean Daily Composite Score Based on the Daytime and Nighttime Asthma Symptom Scores as Measured by Pediatric Asthma Questionnaire
Description: The daily composite score is the sum of the scores of 7 items: Difficulty Breathing, Cough, Wheeze, Activity Limitation, Level of Activity Limitation, Overall Symptom Score, and Nighttime Asthma. The range for the PAQ is 0 (no symptoms) to 27 (severe symptoms).
  The mean daily composite score at Visit 4 is defined as the mean daily composite scores in the 7 days prior to Visit 4.
Time Frame: Baseline, Visit 4 (Week 4)
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 59 | 54
units on a scale | -1.39 (3.213) | -0.91 (2.585) | -0.47 (2.931)

7. Secondary Outcome: Change From Baseline to Visit 2 to Visit 3 in the Mean Daily Composite Score Based on the Daytime and Nighttime Asthma Symptom Scores as Measured by the Pediatric Asthma Questionnaire
Description: The daily composite score is the sum of the scores of 7 items: Difficulty Breathing, Cough, Wheeze, Activity Limitation, Level of Activity Limitation, Overall Symptom Score, and Nighttime Asthma. The range for the PAQ is 0 (no symptoms) to 27 (severe symptoms).
  The mean daily composite score from Visit 2 to Visit 3 is defined as the mean of the daily composite scores from Visit 2 (inclusive) to the day prior to Visit 3.
Time Frame: The days from Visit 2 (inclusive) to the day prior to Visit 3 - approximately 14 days
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 68 | 65 | 59
units on a scale | -0.87 (2.797) | -0.36 (2.872) | -0.08 (2.589)

8. Secondary Outcome: Change From Baseline to Visit 3 to Visit 4 in the Mean Daily Composite Score Based on the Daytime and Nighttime Asthma Symptom Score as Measured by the Pediatric Asthma Questionnaire
Description: The daily composite score is the sum of the scores of 7 items: Difficulty Breathing, Cough, Wheeze, Activity Limitation, Level of Activity Limitation, Overall Symptom Score, and Nighttime Asthma. The range for the PAQ is 0 (no symptoms) to 27 (severe symptoms).
  The mean daily composite score from Visit 3 to Visit 4 is defined as the mean of the daily composite scores from Visit 3 (inclusive) to the day prior to Visit 4.
Time Frame: The days from Visit 3 (inclusive) to the day prior to Visit 4 - approximately 14 days
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 64 | 62 | 57
units on a scale | -1.24 (2.979) | -0.61 (2.706) | -0.37 (2.572)

9. Secondary Outcome: Change From Baseline in In-Clinic Peak Expiratory Flow to Postdose Timepoints at Visit 2
Description: Peak expiratory flow (PEF) measures how fast a person can breathe out using the greatest effort
Time Frame: Baseline, Visit 2: 30 minutes post-dose (on the day of randomization), 1 hour post-dose, 4 hours post-dose, 6 hours post-dose
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 11 | 8 | 8
liters
  Visit 2, 30 minutes post-dose | -0.08 (0.147) | 0.17 (0.211) | 0.16 (0.101)
  Visit 2, 1 hour post-dose | -0.04 (0.183) | 0.13 (0.162) | 0.18 (0.176)
  Visit 2, 4 hours post-dose | -0.09 (0.303) | 0.06 (0.098) | 0.04 (0.188)
  Visit 2, 6 hours post-dose | -0.07 (0.121) | 0.12 (0.164) | 0.06 (0.213)

10. Secondary Outcome: Change From Baseline in In-Clinic Peak Expiratory Flow to Postdose Timepoint at Visit 3
Time Frame: Baseline, Visit 3, pre-dose (approximately 14 days after randomization)
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 11 | 7 | 8
liters | -0.23 (0.255) | 0.14 (0.251) | 0.03 (0.120)

11. Secondary Outcome: Change From Baseline in In-Clinic Peak Expiratory Flow to Postdose Timepoint at Visit 4
Time Frame: Visit 4: pre-dose (approximately 28 days after randomization) , 30 minutes post-dose, 1 hour post-dose, 4 hours post-dose, 6 hours post-dose
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 10 | 7 | 8
liters
  Visit 4, pre-dose | -0.25 (0.307) | 0.29 (0.313) | 0.04 (0.146)
  Visit 4, 30 minutes post-dose | -0.17 (0.323) | 0.29 (0.247) | 0.42 (0.585)
  Visit 4, 1 hour post-dose | -0.03 (0.332) | 0.40 (0.242) | 0.16 (0.227)
  Visit 4, 4 hours post-dose | -0.11 (0.382) | 0.30 (0.305) | 0.11 (0.181)
  Visit 4, 6 hours post-dose | -0.07 (0.260) | 0.20 (0.173) | 0.09 (0.361)

12. Secondary Outcome: Percent Change From Baseline in In-Clinic Peak Expiratory Flow to Postdose Timepoints at Visit 2
Time Frame: Baseline, Visit 2: , 30 minutes post-dose (on the day of randomization), 1 hour post-dose, 4 hours post-dose, 6 hours post-dose
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Levalbuterol UDV: 0.31 ug Levalbuterol UDV TID LEV UDV Levalbuterol UDV TID: 0.31 ug Levalbuterol UDV TID
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 11 | 8 | 8
percent change
  Visit 2, 30 minutes post-does | -5.42 (9.940) | 23.22 (36.195) | 21.71 (23.782)
  Visit 2, 1 hour post-dose | -2.83 (15.094) | 18.21 (26.225) | 25.05 (37.207)
  Visit 2, 4 hours post-dose | -4.22 (17.886) | 9.54 (15.467) | 11.74 (37.114)
  Visit 2, 6 hours post-dose | -5.24 (10.440) | 17.21 (24.013) | 14.40 (41.548)

13. Secondary Outcome: Percent Change From Baseline in In-Clinic Peak Expiratory Flow to Postdose Timepoints at Visit 3
Time Frame: Baseline, Visit 3, pre -dose (approximately 14 days after randomization)
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 11 | 7 | 8
percent change | -18.58 (21.742) | 25.36 (30.129) | 6.02 (13.444)

14. Secondary Outcome: Percent Change From Baseline in In-Clinic Peak Expiratory Flow to Postdose Timepoints at Visit 4
Time Frame: Baseline, Visit 4, pre -dose (approximately 28 days after randomization)
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 10 | 7 | 8
percent change
  Visit 4, pre-dose | -17.26 (23.343) | 49.92 (48.545) | 7.03 (18.829)
  Visit 4, 30 minutes post-dose | -11.69 (27.617) | 48.94 (48.881) | 47.47 (55.010)
  Visit 4, 1 hour post-dose | 0.94 (24.020) | 63.76 (45.620) | 25.32 (47.769)
  Visit 4, 4 hours post-dose | -4.67 (27.435) | 47.59 (42.339) | 20.20 (37.895)
  Visit 4, 6 hours post-dose | -2.06 (21.507) | 32.00 (27.657) | 25.09 (69.440)

15. Secondary Outcome: Change From Baseline in the At-Home Mean Daily Peak Expiratory Flow (PEF to Postdose Timepoint at Visit 3 and Visit 4
Description: Mean of the daily pre-dose PEF values in the week prior to visit in those subjects aged 24 to <48 months capable of performing acceptable and reproducible PEF maneuvers.
Time Frame: Baseline, Visit 3 (the week prior to Visit 3) and Visit 4
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 10 | 8 | 8
liters
  Visit 3 | 0.07 (0.164) | 0.12 (0.209) | 0.01 (0.193)
  Visit 4 | 0.00 (0.205) | 0.08 (0.186) | -0.01 (0.096)

16. Secondary Outcome: Percent Change From Baseline in the At-Home Mean Daily Peak Expiratory Flow (PEF to Postdose Timepoint at Visit 3 and Visit 4)
Description: as for outcome 15
Time Frame: Visit 3 (the week prior to Visit 3), Visit 4 (the week prior to Visit 4)
Population: Intent-to-Treat Population - PEF Cohort (Subjects able to perform PEFs)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 10 | 8 | 8
percent change
  Visit 3 | 7.39 (16.585) | 15.05 (26.849) | 5.30 (21.093)
  Visit 4 | 0.21 (22.426) | 10.33 (24.436) | -1.05 (12.155)

17. Secondary Outcome: Investigator Global Assessment - Question 1
Description: Since the start of the study, how would you evaluate the child's asthma symptoms?
Time Frame: Visit 4 (End of 28 day treatment period)
Population: Intent-to-Treat Population
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 60 | 55
Number of subjects
  Much Better | 12 | 17 | 16
  Moderately Better | 23 | 15 | 13
  Slightly Better | 12 | 14 | 11
  The Same | 14 | 12 | 13
  Slightly Worse | 0 | 1 | 1
  Moderately Worse | 1 | 1 | 1
  Much Worse | 0 | 0 | 0

18. Secondary Outcome: Investigator Global Assessment - Question 2
Description: Since the start of the study, how would you evaluate your ability to manage the subject's asthma?
Time Frame: Visit 4 (End of 28 day treatment period)
Population: Intent-to-Treat Population
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 60 | 55
Number of subjects
  Much Better | 19 | 21 | 23
  Moderately Better | 17 | 12 | 11
  Slightly Better | 8 | 12 | 7
  The Same | 17 | 15 | 14
  Slightly Worse | 0 | 0 | 0
  Moderately Worse | 1 | 0 | 0
  Much Worse | 0 | 0 | 0

19. Secondary Outcome: Caregiver Global Assessment - Question 1
Description: Since the start of the study, how would you evaluate your child's asthma symptoms?
Time Frame: Visit 4 (End of 28 day treatment period)
Population: Intent-to-Treat Population
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 60 | 55
Number of subjects
  Much Better | 21 | 21 | 21
  Moderately Better | 16 | 14 | 13
  Slightly Better | 12 | 12 | 8
  The Same | 12 | 11 | 12
  Slightly Worse | 1 | 2 | 0
  Moderately Worse | 0 | 0 | 1
  Much Worse | 0 | 0 | 0

20. Secondary Outcome: Caregiver Global Assessment - Question 2
Description: Since the start of the study, how would you evaluate your ability to manage your child's asthma?
Time Frame: Visit 4 (End of 28 day treatment period)
Population: Intent-to-Treat Population
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 60 | 55
Number of subjects
  Much Better | 27 | 32 | 29
  Moderately Better | 12 | 6 | 10
  Slightly Better | 11 | 10 | 4
  The Same | 11 | 12 | 12
  Slightly Worse | 1 | 0 | 0
  Moderately Worse | 0 | 0 | 0
  Much Worse | 0 | 0 | 0

21. Secondary Outcome: Caregiver Global Assessment - Question 3
Description: Overall I was: Very satisfied with the control of the child's asthma symptoms while enrolled in this study, Moderately satisfied with the control of the child's asthma symptoms while enrolled in this study, Slightly satisfied with the control of the child's asthma symptoms while enrolled in this study, Not satisfied with the control of the child's asthma symptoms while enrolled in this study or answer Missing
Time Frame: Visit 4 (End of 28 day treatment period)
Population: Intent-to-Treat Population
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 60 | 55
Number of subjects
  Very satisfied | 47 | 45 | 45
  Moderately satisfied | 11 | 12 | 7
  Slightly satisfied | 4 | 2 | 1
  Not satisfied | 0 | 1 | 2

22. Secondary Outcome: Rescue Medication Use: Number of Subjects Using Rescue Medication During the Treatment Period
Description: Number of subjects using rescue medication during the treatment period
Time Frame: Visit 2 to Visit 3 (the first 2 weeks of the study) , Visit 3 to Visit 4 (the second 2 weeks of the study), Visit 2 to Visit 4 (the entire 4 weeks of the study)
Population: Intent-to-Treat Population
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 68 | 65 | 63
Number of subjects
  Visit 2 to Visit 3 the first 2 weeks of the study | 24 | 20 | 14
  Visit 3 to Visit 4 the second 2 weeks of the study | 20 | 20 | 12
  Visit 2 to Visit 4 the entire 4 weeks of the study | 33 | 29 | 20

23. Secondary Outcome: Rescue Medication Use - Change From Baseline in Mean Number of Days Used Per Week When Used
Time Frame: as for outcome 22
Population: Intent-to-Treat Population - Subjects who used rescue medication at any time during the first two weeks of the study and who used rescue medication at any time during baseline
Measure: Mean (Standard Deviation); unit: Days per Week
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 10 | 11 | 3
Days per Week
  Visit 2 to Visit 3 the first 2 weeks of the study | -0.3 (2.43) | -0.8 (2.22) | -1.3 (1.29)
  Visit 3 to Visit 4 the second 2 weeks of the study | -0.8 (1.51) | 0.1 (2.57) | -1.0 (0.94)
  Visit 2 to Visit 4 the entire 4 weeks of the study | -1.1 (1.95) | -0.5 (1.89) | -1.1 (0.73)

24. Secondary Outcome: Rescue Medication Use - Change From Baseline in Mean Number of Doses Used Per Week
Time Frame: as for outcome 22
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Doses per Week
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 68 | 65 | 63
Doses per Week
  Visit 2 to Visit 3 the first 2 weeks of the study | 0.0 (3.14) | 0.1 (2.77) | 0.0 (0.77)
  Visit 3 to Visit 4 the second 2 weeks of the study | -0.4 (3.56) | 0.4 (2.83) | 0.1 (1.28)
  Visit 2 to Visit 4 the entire 4 weeks of the study | -0.2 (3.10) | 0.3 (2.23) | 0.0 (0.96)

25. Secondary Outcome: Rescue Medication Use - Change From Baseline in Mean Number of Doses Used Per Week During Weeks When Used
Time Frame: Visit 2 to Visit 3 (the first 2 weeks of the study), Visit 3 to Visit 4 (the second 2 weeks of the study), Visit 2 to Visit 4 (the entire 4 weeks of the study)
Population: Intent-to-Treat Population - subjects who used rescue medication at any time during the first 2 weeks of the study and who had used rescue medication at any time during baseline
Measure: Mean (Standard Deviation); unit: Doses per Week
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 10 | 11 | 3
Doses per Week
  Visit 2 to Visit 3 the first 2 weeks of the study | -2.1 (8.84) | -0.6 (3.94) | -1.3 (2.08)
  Visit 3 to Visit 4 the second 2 weeks of the study | -2.9 (7.64) | 2.8 (6.27) | -0.8 (1.44)
  Visit 2 to Visit 4 the entire 4 weeks of the study | -2.1 (8.06) | 1.8 (4.75) | -0.8 (1.56)

26. Secondary Outcome: Change From Baseline to Visit 3 and Visit 4 in the Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLA) Composite Score
Description: The PACQLQ composite score was calculated as the mean of the scores of the 13 individual questions. Composite scores could range from 1 to 7. Lower scores indicated greater impact of disease on quality of life.
Time Frame: Visit 3 and Visit 4 (End of 28 day treatment period)
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Number analyzed (Participants) | 62 | 60 | 55
Units on a scale
  Visit 3 | 0.34 (0.888) | 0.35 (0.976) | 0.18 (0.944)
  Visit 4 | 0.41 (0.931) | 0.44 (1.171) | 0.21 (0.883)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: One subject in the randomized to levalbuterol UDV group was not dosed
Arm/Group | Placebo | Levalbuterol MDI | Levalbuterol UDV
Serious Adverse Events (participants affected / at risk) | 0/68 | 1/65 | 3/63
Other Adverse Events (participants affected / at risk) | 28/68 | 31/65 | 27/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=68) | Levalbuterol MDI (N=65) | Levalbuterol UDV (N=63)
Metapneumovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=68) | Levalbuterol MDI (N=65) | Levalbuterol UDV (N=63)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sinusitis Bacterial (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 6 (8) | 2 (2)
Pyrexia (General disorders) | 6 (6) | 3 (3) | 7 (7)
Otitis Media (Infections and infestations) | 5 (6) | 5 (6) | 8 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 5 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish